CLINICAL TRIAL: NCT07070271
Title: Effect of Neurophysiological Facilitation of Respiration on Blood Gases and Duration of Hospitalization in Children With Pneumonia
Brief Title: Effect of Neurophysiological Facilitation of Respiration on Blood Gases and Hospital Stay in Children With Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asmaa Ahmed Abd El-samad (Other)
Responsible Party: Sponsor-Investigator, Asmaa Ahmed Abd El-samad, Principal Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005586
Record Dates: First submitted 2025-07-01; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pneumonia
Keywords: Pneumonia; Neurophysiological facilitation; Chest physical therapy; Blood gases
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional chest physical therapy (Active Comparator): Children in this group will only receive conventional chest physical therapy program in form of (postural drainage, chest percussion, vibration and suction if needed).
  Interventions: Other: conventional chest physical therapy
- Conventional chest physical therapy + Neurophysiological facilitation techniques (Experimental): Children in this group will receive conventional chest physical therapy program along with respiratory neurophysiological facilitation techniques in form of (anterior basal lift, intercostal stretch, abdominal co-contraction).
  Interventions: Other: Respiratory neurophysiological facilitation techniques; Other: conventional chest physical therapy

INTERVENTIONS:
Other: Respiratory neurophysiological facilitation techniques — The respiratory neurophysiological facilitation techniques in form of (anterior basal lift, intercostal stretch, abdominal co-contraction) once a day for 5 days.
  Arms: Conventional chest physical therapy + Neurophysiological facilitation techniques
Other: conventional chest physical therapy — conventional chest physical therapy program in form of (postural drainage, chest percussion, vibration and suction if needed) once a day for 5 days.

SUMMARY:
The goal of this clinical trial is to investigate the effect of respiratory neurophysiological facilitation techniques on arterial blood gases, the severity of respiratory illness and duration of hospital stay in hospitalized children with pneumonia.

DETAILED DESCRIPTION:
Children who were hospitalized with a clinically and radiologically confirmed diagnosis of pneumonia will participate in this study. Selected Patients will be randomly assigned into two groups of equal number.

One group will only receive conventional chest physical therapy program in form of (postural drainage, chest percussion, vibration and suction if needed). The other group will receive conventional chest physical therapy program along with respiratory neurophysiological facilitation techniques in form of (anterior basal lift, intercostal stretch, abdominal co-contraction).

All patients will receive the treatment program once a day for successive 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes, with age ranged from 6 months to 2 years old.
* All children diagnosed with pneumonia.
* All children should be vitally stable during the study period.

Exclusion Criteria:

* Medically unstable children.
* Children with uncontrolled convulsions.
* Children with Osteopenia.

Ages: 6 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Arterial blood gases | At baseline (after enrollment and before the first chest physiotherapy session) and on day 5 after completing the fifth session, assessed within 5 days of enrollment
  Blood gas analysis is a commonly used diagnostic tool to evaluate the partial pressures of gas in blood and acid-base content.
  The blood sample is collected from the radial artery or the femoral artery.
Duration of hospitalization | From the date of hospital admission until the date of discharge, up to 20 days
The severity of respiratory illness. | At baseline (after enrollment and before the first chest physiotherapy session) and on day 5 after completing the fifth session, assessed within 5 days of enrollment
  Using the Pediatric Respiratory Severity Score to assess respiratory rate, wheezing, accessory muscle use, SpO2, and feeding difficulties.
  Each component was given 0 or 1 point and the total score was classified as mild (0-1 points), moderate (2-3 points), or severe (4-5 points)

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa Ahmed Abd El-samad, master's degree, Principal Investigator — Cairo University
Locations (1):
- Cairo university specialized pediatric hospital (Abo-El Reesh), Giza, Egypt

IPD SHARING:
Plan to Share IPD: No